CLINICAL TRIAL: NCT05024669
Title: Efficacy of Three Commercially Available Desensitizers in Reducing Post-operative Sensitivity Following Composite Restorations: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Desensitizers in Reducing Post-operative Sensitivity Following Composite Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Dr Harisha Dewan, Assistant Professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Harisha
Record Dates: First submitted 2021-08-14; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Sensitivity
Keywords: Gluma; Sheildforce Plus; Telio CS; Desensitisers
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control Group (No Intervention): where no desensitizer application was done,
- Group GL (Experimental): applied with Gluma dentin desensitizer
  Interventions: Combination Product: Gluma desensitiser
- Group SF (Experimental): applied with Shieldforce desensitizer
  Interventions: Combination Product: Sheildforce Plus desensitiser
- Group TC (Experimental): applied with Telio CS desensitizer
  Interventions: Combination Product: Telio CS desensitiser

INTERVENTIONS:
Combination Product: Gluma desensitiser — Gluma desensitiser was used before restoration.
  Arms: Group GL
Combination Product: Sheildforce Plus desensitiser — Sheildforce Plus desensitiser was used before restoration.
  Arms: Group SF
Combination Product: Telio CS desensitiser — Telio CS desensitiser was used before restoration.
  Arms: Group TC

SUMMARY:
Composite is one of the common aesthetic restorations used in the dentistry. With the advancements in the biomaterials the application of the composites has broadened. However due to various factors the composites are associated with dental sensitivity. Hence in our study we evaluate and compare the effectiveness of three desensitizing agents in reducing the post-treatment sensitivity for class I composite restoration.

DETAILED DESCRIPTION:
A double-blind, randomized, controlled clinical trial was conducted in which 80 subjects requiring class I cavity were randomly assigned to 4 groups of 20 patients each: Group C (Control group), Group GL (Gluma group), Group SF (Shield Force Plus group), and Group TC (Telio CS group). The class 1 cavity was prepared and after etching, the desensitizers were applied (except in the control group) and later composite restoration was done. The postoperative pain/sensitivity level was recorded according to the Visual Analogue Scale (VAS) on intake of cold drinks; intake of hot drinks; and intake of sugar for different periods of time.

ELIGIBILITY:
Inclusion Criteria:

The selection criteria:

* Age was 20-45 years.
* Vital teeth, (electric pulp test)
* Apical periodontal ligament space radiographically identified
* The remaining dentin thickness at least 1mm.

Exclusion Criteria:

* Restored, periodontally weak nonvital teeth are excluded.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Effect of application of the desensitisers on post operative sensitivity on the day of composite restoration on application of different stimuli like (i) Intake of cold drinks; (ii) Intake of hot drinks; and (iii) Intake of sugar. | Within 24 hours
  The patients were given a questionnaire and instructed to record any postoperative pain/sensitivity level according to the Visual Analogue Scale (VAS) for restored tooth on the day of restoration on taking cold drinks, hot drinks, and sugar.
Effect of application of the desensitisers on post operative sensitivity one week after the composite restoration on application of different stimuli like (i) Intake of cold drinks; (ii) Intake of hot drinks; and (iii) Intake of sugar. | After one week
  The patients were given a questionnaire and instructed to record any postoperative pain/sensitivity level according to the Visual Analogue Scale (VAS) for restored tooth one week after the restoration on taking cold drinks, hot drinks, and sugar.
Effect of application of the desensitisers on post operative sensitivity one month after the composite restoration on application of different stimuli like (i) Intake of cold drinks; (ii) Intake of hot drinks; and (iii) Intake of sugar. | after one month
  The patients were given a questionnaire and instructed to record any postoperative pain/sensitivity level according to the Visual Analogue Scale (VAS) for restored tooth one month after the restoration on taking cold drinks, hot drinks, and sugar.

CONTACTS AND LOCATIONS:
Overall Officials: Harisha Dewan, Principal Investigator — University of Jazan
Locations (1):
- Harisha Dewan, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
no plan